CLINICAL TRIAL: NCT00617734
Title: A Randomized Phase 2 Open-Label Study of IMC-A12, as a Single Agent or in Combination With Cetuximab, in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck and Disease Progression on Prior Platinum-Based Chemotherapy
Brief Title: Study of IMC-A12, Alone or in Combination With Cetuximab, in Participants With Recurrent or Metastatic Squamous Cell Carcinoma (MSCC) of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13913; CP13-0706 (Other: ImClone, LLC); CP02-0758 (Other: ImClone, LLC); I5A-IE-JAEB (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-01-30; First posted 2008-02-18 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Cancer
Keywords: Squamous Cell Carcinoma in Head and Neck; Prior Platinum-based chemotherapy; Cetuximab; Erbitux; IMC-A12
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — cixutumumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMC-A12 (cixutumumab) (Experimental)
  Interventions: Biological: IMC-A12 (cixutumumab)
- IMC-A12 (cixutumumab) + cetuximab (Experimental)
  Interventions: Biological: IMC-A12 (cixutumumab); Biological: cetuximab (Erbitux ®)

INTERVENTIONS:
Biological: IMC-A12 (cixutumumab) — IMC-A12 10 milligrams per kilogram (mg/kg) over one hour every two weeks. A cycle is defined as four weeks of therapy. Participants will continue on study until evidence of progressive disease, or unacceptable toxicity develops.
  Other Names: Cixutumumab; LY3012217
Biological: cetuximab (Erbitux ®) — IMC-A12 10 mg/kg over one hour followed by cetuximab 500 milligrams per square meter (mg/m^2) over two hours. This sequence will be repeated every two weeks. Participants will continue on study until evidence of progressive disease or unacceptable toxicity develops.
  Other Names: Erbitux®
  Arms: IMC-A12 (cixutumumab) + cetuximab

SUMMARY:
The purpose of this study is to determine if IMC-A12 alone or in combination with Cetuximab (Erbitux®) can increase the time prior to disease progression in participants with Squamous Cell Head and Neck Cancer who have had disease progression and platinum-containing chemotherapeutic regimen.

DETAILED DESCRIPTION:
The routine cancer treatments for Squamous Cell Carcinoma Head and Neck Cancer have improved but still leave a percentage of participants with incurable disease. New alternatives for participants whose disease is refractory to existing therapies is needed.

IMC-A12 is a monoclonal antibody which binds to special receptors known as insulin-like growth factor-I receptor (IGF-IR). This binding action has been shown to inhibit the growth of a variety of human tumor cell lines.

The purpose of this study is to evaluate the effects of IMC-A12 by itself or with Cetuximab (Erbitux®) in participants with Squamous Cell Carcinoma Head and Neck Cancer that has spread to other parts of the body, and to determine how long the drug remains in the body. The study will also look at what side effects IMC-A12 may cause when a participant is receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed squamous cell carcinoma of the oropharynx, hypopharynx, larynx, or oral cavity, metastasis or recurrence documented by clinical imaging studies
* Measurable disease, lesion size ≥ 2 centimeters (cm) on conventional measurement techniques or ≥ 1 cm on spiral computed tomography (CT) scan
* Clinical documentation of disease progression during treatment with or within 90 days after receiving the last cycle of platinum-based chemotherapy (with or without radiation therapy)
* If prior treatment with anti-epidermal growth factor receptor (EGFR) therapy, the time to recurrence from last exposure to anti-EGFR therapy is > 90 days
* Adequate hematologic function
* Adequate hepatic function
* Adequate coagulation function or is on a stable dose of an anticoagulant.
* Adequate renal function
* Fasting serum glucose <120 milligrams per deciliter (mg/dL) or below the upper limit of normal (ULN)
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

Exclusion Criteria:

* Not recovered from adverse events due to agents administered more than 4 weeks earlier. Neurotoxicity, must have recovered to grade ≤ 2
* Is receiving any other investigational agent(s)
* History of treatment with other agents targeting the insulin-like growth factor receptor (IGFR)
* Is receiving concurrent treatment with other anticancer therapy, including chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemoembolization, or targeted therapy
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab or IMC-A12
* Has poorly controlled diabetes mellitus. Participants with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within normal range (fasting < 120 mg/dL or below ULN) and that they are on a stable dietary or therapeutic regimen for this condition
* Pregnant or breastfeeding
* Is receiving therapy with immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-03; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (14):
  - ImClone Investigational Site, Orange, California
  - ImClone Investigational Site, Miami, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Baltimore, Maryland
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Rochester, Minnesota
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, The Bronx, New York
  - ImClone Investigational Site, Pittsburgh, Pennsylvania
  - ImClone Investigational Site, Nashville, Tennessee
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Presented are the reasons the participants discontinued from the study treatment.
Groups:
- IMC-A12 (Cixutumumab): IMC-A12 (cixutumumab) 10 milligrams per kilogram (mg/kg) dose administered as an intravenous (IV) infusion over a period of 1 hour once every 2 weeks. A cycle was defined as 4 weeks of therapy. (4-week cycle). Treatment was continued until there was evidence of progressive disease (PD), unacceptable toxicity, or withdrawal of consent.
- IMC-A12 (Cixutumumab) + Cetuximab: IMC-A12 (cixutumumab) 10 mg/kg dose administered as an IV infusion over a period of 1 hour followed by cetuximab 500 milligrams per square meter (mg/m^2) administered as an IV infusion over a period of 2 hours; this sequence was repeated once every 2 weeks (4-week cycle). Treatment was continued until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Started | 49 | 48
Received at Least 1 Dose of Study Drug | 47 | 44
Completed | 41 | 42
Not Completed | 8 | 6
Not completed — Withdrew Consent | 2 | 0
Not completed — Adverse Event | 4 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Found Ineligible After Randomization | 1 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug.
Groups:
- IMC-A12 (Cixutumumab): IMC-A12 (cixutumumab) 10 mg/kg dose administered as an IV infusion over a period of 1 hour once every 2 weeks. A cycle was defined as 4 weeks of therapy (4-week cycle). Treatment was continued until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
- IMC-A12 (Cixutumumab) + Cetuximab: IMC-A12 (cixutumumab) 10 mg/kg dose administered as an IV infusion over a period of 1 hour followed by cetuximab 500 mg/m^2 dose administered as an IV infusion over a period of 2 hours; this sequence was repeated once every 2 weeks (4-week cycle). Treatment was continued until there was evidence of PD, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab | Total
Number analyzed (Participants) | 47 | 44 | 91
Age, Continuous [Median (Full Range); unit: years] | 60.0 [46.0 to 81.0] | 59.0 [35.0 to 76.0] | 60.0 [35.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 36 | 37 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 46 | 40 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 34 | 76
  Black or African American | 3 | 5 | 8
  Asian | 0 | 2 | 2
  Other | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 44 | 91
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 171.7 (10.53) | 173.3 (9.56) | 172.5 (10.05)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 70.5 (13.68) | 70.9 (18.19) | 70.7 (15.93)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meters (m^2)] — BSA is the measured or calculated surface area of a human body based on body weight and height.
  The Mosteller¹ formula to calculate BSA (m^2) = ([Height (centimeter) x Weight (kilograms)]/ 3600)½.
  square meters (m^2) | 1.80 (0.241) | 1.82 (0.269) | 1.81 (0.254)
Electrocardiogram (ECG) [Count of Participants; unit: Participants]
  Normal | 20 | 26 | 46
  Abnormal | 27 | 18 | 45
Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score [Count of Participants; unit: Participants] — ECOG performance status was used to classify participants according to their functional impairment. Score 0 = Fully active, able to carry on all pre-disease performance without restriction. Score 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, for example, light house work, office work. Score 2 = Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 = Fully Active | 8 | 8 | 16
    1 = Ambulatory, Restricted Work Activity | 29 | 28 | 57
    2 = Ambulatory, No Work Activity | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the interval from randomization until PD or death, whichever occurred first. Response was defined using Response Evaluation Criteria in Solid Tumors (RECIST, version 1.0) criteria. PD was defined as having at least a 20% increase in sum of the longest diameter of target lesions or the appearance of new lesions. PFS was censored at the date of the last objective progression-free disease assessment for participants who did not experience PD or death.
Time Frame: Baseline to measured PD (up to 27.66 months)
Population: Randomized participants who received at least 1 dose of study drug. Seven (7) participants in IMC-A12 (Cixutumumab) and 4 participants in IMC-A12 (Cixutumumab) + Cetuximab were censored for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Number analyzed (Participants) | 47 | 44
months | 1.9 [1.6 to 1.9] | 2.0 [1.8 to 3.5]
Statistical Analysis 1: Comparison: IMC-A12 (Cixutumumab) vs IMC-A12 (Cixutumumab) + Cetuximab; Test type: Superiority or Other; p = 0.0667, Log Rank

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: ORR was defined as the percentage of participants achieving either CR or PR. Response was defined using RECIST, version 1.0 criteria. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Percentage of participants is calculated as a total number of participants with CR or PR divided by the total number of participants treated then multiplied by 100.
Time Frame: Baseline to measured PD (up to 27.66 months)
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Number analyzed (Participants) | 47 | 44
percentage of participants | 2.1 [0.1 to 9.7] | 9.1 [3.2 to 19.6]
Statistical Analysis 1: Comparison: IMC-A12 (Cixutumumab) vs IMC-A12 (Cixutumumab) + Cetuximab; Test type: Superiority or Other; p = 0.1935, Fisher Exact

3. Secondary Outcome: Percentage of Participants With PFS at 6 Months
Description: PFS at 6 months was defined as the percentage of participants who have neither experienced PD nor died at 6 months after the date of randomization. Response was defined using RECIST, version 1.0 criteria. PD was defined as having at least a 20% increase in sum of the longest diameter of target lesions or the appearance of new lesions. Percentage of participants is calculated as the total number of participants with PFS at 6 months divided by the total number of participants treated then multiplied by 100.
Time Frame: 6 months
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Number analyzed (Participants) | 47 | 44
percentage of participants | 4.3 [0.5 to 14.5] | 13.6 [5.2 to 27.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from the date of randomization to the date of death from any cause. For participants who were alive, OS was censored at the date of last follow-up visit or at the date of last contact.
Time Frame: Baseline to date of death from any cause (up to 29.63 months)
Population: Randomized participants who received at least 1 dose of study drug. Eleven (11) participants in IMC-A12 (Cixutumumab) group and 6 participants in IMC-A12 (Cixutumumab) + Cetuximab group were censored for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Number analyzed (Participants) | 47 | 44
months | 5.3 [4.3 to 8.0] | 5.5 [4.3 to 7.4]
Statistical Analysis 1: Comparison: IMC-A12 (Cixutumumab) vs IMC-A12 (Cixutumumab) + Cetuximab; Test type: Superiority or Other; p = 0.7455, Log Rank

5. Secondary Outcome: Duration of Response
Description: The duration of CR or PR was defined as the time from first objective status assessment of CR or PR to the first time of PD or death. Response was defined using RECIST, version 1.0 criteria. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Duration of response was censored on the date of last tumor assessment for participants who were alive and have no evidence of PD.
Time Frame: Date of first response to the date of PD or death due to any cause (up to 23.98 months)
Population: Randomized participants who received at least 1 dose of study drug and had CR or PR. No participants were censored for duration of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Number analyzed (Participants) | 1 | 4
months | 12.8 [NA to NA] — 95% confidence interval was not estimable as only one participant had response. | 6.2 [3.58 to 23.98]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Deaths
Description: TEAEs were defined as serious and other non-serious adverse events (AEs) that occurred or worsened after study treatment (regardless of causality). Data presented are the number of participants who experienced TEAEs including serious TEAEs, and deaths during the study including the 30-day follow-up. A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events section of this report.
Time Frame: Baseline through study completion (up to 29.63 months)
Population: Randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Number analyzed (Participants) | 47 | 44
participants
  TEAEs | 47 | 44
  Serious TEAEs | 20 | 23
  Death due to AEs | 2 | 6

7. Secondary Outcome: Blood And Tissue Biomarkers And Development of Serum Antibodies Against IMC-A12 and Cetuximab
Description: No data for biomarkers and serum antibodies were collected due to lack of an appropriate validated assay.
Time Frame: Biomarkers [pre-dose, Cycle 1 (Day 15), (Cycle 2 (Day 1), and end of treatment]; Immunogenicity [pre-dose, prior to first infusion for Cycle 3, Cycle 5, and 30-day safety follow-up]
Population: No participants were analyzed due to lack of an appropriate validated assay.
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | IMC-A12 (Cixutumumab) | IMC-A12 (Cixutumumab) + Cetuximab
Serious Adverse Events (participants affected / at risk) | 20/47 | 23/44
Other Adverse Events (participants affected / at risk) | 44/47 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 (Cixutumumab) (N=47) | IMC-A12 (Cixutumumab) + Cetuximab (N=44)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Scotoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (6)
Oral cavity fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (6)
Asthenia (General disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 2 (2) | 3 (3)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 6 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Gastrostomy tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 (Cixutumumab) (N=47) | IMC-A12 (Cixutumumab) + Cetuximab (N=44)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (5)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 5 (6)
Dry eye (Eye disorders) | 3 (3) | 2 (2)
Breath odour (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 9 (14)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 13 (16) | 13 (17)
Oral pain (Gastrointestinal disorders) | 4 (4) | 6 (8)
Salivary gland disorder (Gastrointestinal disorders) | 3 (3) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 13 (18)
Vomiting (Gastrointestinal disorders) | 9 (10) | 7 (11)
Fatigue (General disorders) | 26 (35) | 27 (35)
Oedema (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 7 (8)
Candidiasis (Infections and infestations) | 3 (3) | 3 (7)
Localised infection (Infections and infestations) | 0 (0) | 3 (6)
Oral infection (Infections and infestations) | 3 (3) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 8 (10)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Weight decreased (Investigations) | 12 (13) | 13 (18)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 8 (11)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (16) | 13 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 6 (8)
Dysarthria (Nervous system disorders) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 8 (9) | 11 (11)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 28 (46)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (8)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (8)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Haemorrhage (Vascular disorders) | 3 (5) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.